CLINICAL TRIAL: NCT06680544
Title: Comparing the Efficacy of Oral 200 Milligram Voriconazole Once a Day Vs. Twice a Day in the Treatment of Resisitant Dermatophyte Infections (Tinea Corporis and Tinea Cruris)
Brief Title: Role of Oral Voriconazole in the Treatment of Resistant Dermatophyte Infections
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Muhammad Khurram Shahzad, Senior Registrar Dermatology, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZMC/H
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Dermatophyte Infection
Keywords: Tinea; Voriconazole; Dermatomycoses; Antifungal Agents
MeSH Terms: conditions — Dermatomycoses; Tinea | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oral voriconazole 200 mg once daily group (group A) (Active Comparator): Patients with resistant dermatophyte infection (tinea corporis and cruris)will be given oral voriconazole 200 mg once daily
  Interventions: Drug: Voriconazole low dose
- oral voriconazole 200 mg twice daily group (group B) (Active Comparator): Patients with resistant dermatophyte infection (tinea corporis and cruris)will be given oral voriconazole 200 mg twice daily
  Interventions: Drug: Voriconazole high dose

INTERVENTIONS:
Drug: Voriconazole high dose — Oral voriconazole 200mg once a day for a maximum of 28 days
  Arms: oral voriconazole 200 mg twice daily group (group B)
Drug: Voriconazole low dose — Oral voriconazole 200mg twice a day for a maximum of 28 days
  Arms: oral voriconazole 200 mg once daily group (group A)

SUMMARY:
Treatment of dermatophyte infection in our country (Pakistan) is becoming difficult due to the developing resistance to traditional antifungal agents. Assessing the effectiveness ,feasibility and standard dosage of a newer antifungal drug like voriconazole is the need of the hour in resistant cases of dermatophyte infection.

DETAILED DESCRIPTION:
Treatment of dermatophyte infection in our country is becoming difficult due to the developing resistance to traditional antifungal agents. Assessing the effectiveness and feasibility of a newer antifungal drug like voriconazole is the need of the hour in resistant cases.

Objective: To compare the efficacy of oral 200 milligram voriconazole once a day vs twice a day in the treatment of resistant dermatophyte infections (tinea corporis and cruris).

Material & Methods: This randomized controlled trial using non-probability sampling technique will be carried out in Outpatient Dermatology Department, Sheikh Zayed Hospital Rahim Yar Khan, Pakistan. Approval from ethical review committee of the hospital has been taken. Total 106 patients will be divided into two groups, Group A and Group B, each consisting of 53 patients. Group A will be given oral voriconazole 200mg once a day and Group B will be given twice a day for a maximum of 28 days. Efficacy will be assessed at day 14 and day 28, and relapse will be noted at the 2-month follow-up visit. Data will be recorded on a preformed Proforma for each patient and wiil be analyzed using SPSS 24. A p-value of less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Resistant cases of tinea cruris and tinea corporis: Those cases who received the standard dosage of oral antifungals i.e. oral terbinafine 5mg/kg per day for 4 weeks or oral itraconazole 5mg per/kg/day for 4 weeks but they did not recover from the infection.
2. Skin area: Groin and trunk
3. Total diameter of the lesions: 5cm to 80 cm

Exclusion Criteria:

1. History of hypersensitivity to azoles
2. All those individuals having immunocompromised state (malignancy, tuberculosis, AIDS, history of organ transplant and history of immunosuppressive drug treatment etc.)
3. Patients of diabetes, liver or kidney disease.
4. Lactating mother
5. Pregnant female

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy of oral voriconazole 200 mg once daily(low dose) vs. twice daily (high dose) | Clinical assessment for efficacy will be done at day 14 and day 28
  Efficacy will be assesssed clinically either through complete resolution of lesion or leaving behind pigmentation

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh zayed Medical College and Hospital, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No